CLINICAL TRIAL: NCT00819013
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Safety, Reactogenicity, and Immunogenicity of Recombinant M2e Influenza-A Vaccine Candidate ACAM FLU-A) in Healthy Adults
Brief Title: Safety Study of Recombinant M2e Influenza-A Vaccine in Healthy Adults
Acronym: FLU-A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-261-001
Record Dates: First submitted 2008-10-10; First posted 2009-01-08 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study Group 1 (Experimental): ACAM-FLU-A low dose + Adjuvant 1
  Interventions: Biological: Influenza A Vaccine: ACAM FLU-A
- Study Group 2 (Experimental): ACAM-FLU-A low dose + Adjuvant 2
  Interventions: Biological: Influenza A Vaccine: ACAM FLU-A
- Study Group 3 (Experimental): ACAM-FLU-A low dose
  Interventions: Biological: Influenza A Vaccine: ACAM FLU-A
- Study Group 4 (Placebo Comparator): Saline placebo
  Interventions: Biological: Saline placebo

INTERVENTIONS:
Biological: Influenza A Vaccine: ACAM FLU-A — 0.5 mL ACAM-FLU-A low dose + Adjuvant 1, Intramuscular
  Other Names: ACAM FLU-A
  Arms: Study Group 1
Biological: Influenza A Vaccine: ACAM FLU-A — 0.5 mL ACAM-FLU-A low dose + Adjuvant 2, Intramuscular
  Other Names: ACAM FLU-A
  Arms: Study Group 2
Biological: Influenza A Vaccine: ACAM FLU-A — 0.5 mL ACAM FLU-A low dose, Intramuscular
  Other Names: ACAM FLU-A
  Arms: Study Group 3
Biological: Saline placebo — 0.5 mL, Intramuscular
  Other Names: USP Saline
  Arms: Study Group 4

SUMMARY:
This multi-center study will be conducted in the United States with up to 80 healthy adult subjects. Subjects will be scheduled to receive a total of two (2) injections with 1 injection each administered.

Subjects will be randomized according to a randomization scheme.

DETAILED DESCRIPTION:
All subjects will be followed up for 60 days post-randomization and through the influenza season. Following the influenza season, a subset of the subjects will receive a booster vaccine at the 12 month time point. The subjects will further be assessed at 2 days, 7 days, 15 days, 30 days and 6 months following the booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females 18 - 40 years of age in good general health

Exclusion Criteria:

* Known allergies or severe reactions to any of the vaccine components including those to adjuvants
* History of severe allergic reactions, including angioedema;
* History of asthma or recurrent wheezing; (current or within past 2 years);
* History of neurological symptoms or signs following administration of any vaccine;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (3):
- United States (3):
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Northwest Kinetics, Tacoma, Washington

REFERENCES:
- [Derived] Ibanez LI, Roose K, De Filette M, Schotsaert M, De Sloovere J, Roels S, Pollard C, Schepens B, Grooten J, Fiers W, Saelens X. M2e-displaying virus-like particles with associated RNA promote T helper 1 type adaptive immunity against influenza A. PLoS One. 2013;8(3):e59081. doi: 10.1371/journal.pone.0059081. Epub 2013 Mar 18. PMID 23527091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 11 to 27 July 2007 at 3 clinical centers in the US.
Pre-assignment Details: A total of 87 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- ACAM-FLU-A Adjuvanted With Alhydrogel: Participants who received a 0.5 mL dose of ACAM FLU A vaccine adjuvanted with Alhydrogel, on Day 0 and Day 30.
- ACAM-FLU-A Adjuvanted With Stimulon® QS-21: Participants who received a 0.5 mL dose of ACAM FLU A vaccine adjuvanted with Stimulon QS 21, on Day 0 and Day 30.
- ACAM FLU A Without Adjuvant: Participants who received 0.5 mL dose of ACAM FLU A vaccine without adjuvant, on Day 0 and Day 30.
- Saline Placebo: Participants who received a 0.5 mL dose of placebo (saline) vaccine, on Day 0 and Day 30.
Period: Overall Study
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Started | 22 | 23 | 21 | 21
Completed | 19 | 22 | 16 | 17
Not Completed | 3 | 1 | 5 | 4
Not completed — Not meeting continuing study eligibility | 2 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo | Total
Number analyzed (Participants) | 22 | 23 | 21 | 21 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 21 | 21 | 87
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (5.91) | 27.7 (4.96) | 27.9 (6.76) | 29.4 (6.84) | 28.5 (6.1175)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 10 | 10 | 39
  Male | 15 | 11 | 11 | 11 | 48
Region of Enrollment [Number; unit: Participants]
  United States | 22 | 23 | 21 | 21 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events by System Organ Class After Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or a Placebo Vaccine.
Time Frame: Day 0 through Day 60 post-vaccination
Population: Safety assessments were on participants who received the initial injection and had at least one post-baseline immunogenicity assessment, regardless of the time of follow-up or protocol deviations - Intent to Treat Population.
Measure: Number; unit: Participants
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 22 | 23 | 21 | 21
Participants
  Blood and Lymphatic System Disorders | 2 | 2 | 1 | 0
  Cardiac Disorders | 0 | 1 | 0 | 0
  Ear and Labyrinth Disorders | 0 | 0 | 0 | 1
  Eye Disorders | 1 | 0 | 0 | 0
  Gastrointestinal Disorders | 4 | 7 | 4 | 5
  General and Administration Site Disorders | 21 | 22 | 18 | 10
  Hepatobiliary Disorders | 0 | 1 | 0 | 0
  Immune System Disorders | 1 | 0 | 0 | 0
  Infections and Infestations | 3 | 2 | 4 | 4
  Injury, Poisoning and Procedural Complications | 1 | 1 | 0 | 1
  Investigations | 17 | 19 | 20 | 15
  Musculoskeletal and Connective Disorders | 6 | 12 | 8 | 4
  Neoplasms Benign, Malignant, and Unspecified | 1 | 0 | 1 | 0
  Nervous System Disorders | 8 | 12 | 6 | 3
  Psychiatric Disorders | 0 | 0 | 1 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 4 | 5 | 8 | 5
  Skin and Subcutaneous Tissue Disorders | 1 | 0 | 1 | 1

2. Primary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Adverse Event After Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Description: Solicited Injection Site Adverse Events: Erythema, Induration, Pain, Pruritus, Swelling, Rash. Solicited Systemic Adverse Events: Lymph Node Pain, Pyrexia (Temperature), Chills, Constipation, Diarrhoea, Fatigue, Headache, Malaise, Myalgia, Nausea, Vomiting, Alanine Aminotransferase Increased, Aspartate Aminotransferase Increased, Blood Creatinine Increased, Haemoglobin Decreased, Platelet Count Decreased, White Blood Cell Count Increased.
Time Frame: Day 0 through Day 7 post-vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 22 | 23 | 21 | 21
Participants
  Lymph Node Pain (Post-dose 1) | 1 | 0 | 1 | 0
  Pyrexia (Temperature; [Post-dose 1]) | 3 | 3 | 0 | 1
  Chills (Post-dose 1) | 0 | 2 | 0 | 1
  Constipation (Post-dose 1) | 0 | 0 | 0 | 1
  Diarrhoea (Post-dose 1) | 2 | 0 | 1 | 2
  Fatigue Post (Post-dose 1) | 4 | 6 | 1 | 3
  Headache (Post-dose 1) | 4 | 6 | 1 | 0
  Malaise (Post-dose 1) | 1 | 3 | 1 | 1
  Myalgia (Post-dose 1) | 5 | 8 | 1 | 2
  Nausea (Post-dose 1) | 0 | 0 | 0 | 1
  Alanine Aminotranferase Increased (Post-dose 1) | 1 | 0 | 1 | 0
  Blood Creatinine Increased (Post-dose 1) | 0 | 1 | 0 | 0
  Haemoglobin Decreased (Post-dose 1) | 3 | 5 | 1 | 4
  Platelet Count Decreased (Post-dose 1) | 1 | 0 | 0 | 0
  White Blood Cell Count Increased (Post-dose 1) | 0 | 1 | 0 | 1
  Injection Site Erythema (Post-dose 1) | 0 | 1 | 2 | 0
  Injection Site Pain (Post-dose 1) | 14 | 18 | 12 | 1
  Injection Site Pruritus (Post-dose 1) | 0 | 2 | 1 | 2
  Injection Site Swelling (Post-dose 1) | 1 | 4 | 0 | 0
  Pyrexia (Temperature; [Post-dose 2]) | 1 | 9 | 2 | 1
  Chills (Post-dose 2) | 0 | 6 | 0 | 1
  Diarrhoea (Post-dose 2) | 0 | 1 | 0 | 0
  Fatigue (Post-dose 2) | 2 | 8 | 0 | 1
  Headache (Post-dose 2) | 1 | 6 | 1 | 1
  Malaise (Post-dose 2) | 2 | 8 | 0 | 1
  Myalgia (Post-dose 2) | 1 | 8 | 1 | 1
  Nausea (Post-dose 2) | 0 | 3 | 0 | 1
  Vomiting (Post-dose 2) | 0 | 0 | 0 | 1
  Alanine Aminotranferase Increased (Post-dose 2) | 1 | 1 | 1 | 0
  Aspartate Aminotranferase Increased (Post-dose 2) | 0 | 1 | 0 | 0
  Haemoglobin Decreased (Post-dose 2) | 0 | 1 | 1 | 0
  Platelet Count Decreased Post Dose 2 | 1 | 0 | 0 | 0
  White Blood Cell Count Increased (Post-dose 2) | 0 | 1 | 0 | 0
  Injection Site Erythema (Post-dose 2) | 3 | 6 | 3 | 2
  Injection Site Induration (Post-dose 2) | 2 | 1 | 3 | 0
  Injection Site Pain (Post-dose 2) | 12 | 17 | 7 | 2
  Injection Site Pruritus (Post-dose 2) | 0 | 1 | 0 | 0
  Injection Site Swelling (Post-dose 2) | 1 | 4 | 0 | 0
  Injection Site Rash (Post-dose 2) | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Evaluated Laboratory Abnormalities After Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Time Frame: Day 0 through Day 60 post-vaccination 1
Population: Laboratory parameters were assessed in participants who received the initial injection and had at least one post-baseline immunogenicity assessment, regardless of the time of follow-up or protocol deviations (Intent-to-treat Population).
Measure: Number; unit: Participants
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 22 | 23 | 21 | 21
Participants
  Alanine Aminotranferase Increase | 1 | 2 | 2 | 1
  Aspartate Aminotransferase Increase | 0 | 3 | 0 | 0
  Blood Bilirubin Decreased | 2 | 7 | 7 | 3
  Blood Bilirubin Increased | 0 | 3 | 0 | 0
  Blood Creatine Increased | 0 | 1 | 0 | 0
  Blood Creatine Phosphokinase Increased | 6 | 5 | 3 | 4
  Blood Creatinine Decreased | 0 | 0 | 0 | 1
  Blood Creatinine Increased | 6 | 4 | 6 | 4
  Blood Glucose Decreased | 0 | 2 | 0 | 0
  Blood Glucose Increased | 2 | 3 | 3 | 3
  Blood Potassium Increased | 3 | 2 | 3 | 1
  Blood Urea Increased | 1 | 0 | 0 | 0
  Blood Urine | 0 | 0 | 0 | 1
  Eosinophil Count Increased | 0 | 0 | 1 | 0
  Glucose Urine | 0 | 0 | 0 | 1
  Haemoglobin Decreased | 7 | 8 | 7 | 5
  Lymphocyte Count Decreased | 0 | 2 | 1 | 0
  Lymphocyte Count Increased | 0 | 0 | 1 | 0
  Nitrite Urine Present | 0 | 0 | 0 | 1
  Platelet Count Decreased | 1 | 0 | 0 | 0
  Platelet Count Increased | 0 | 1 | 1 | 1
  Protein Urine Present | 2 | 3 | 1 | 1
  Red Blood Cells Urine | 0 | 1 | 2 | 1
  Urine Leukocyte Esterase Positive | 0 | 1 | 0 | 2
  White Blood Cell Count Decreased | 2 | 3 | 1 | 1
  White Blood Cell Count Increased | 0 | 2 | 1 | 2
  White Blood Cells Urine | 0 | 1 | 0 | 2

4. Secondary Outcome: Number of Participants With Signs and Symptoms of Influenza After Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Description: Participants who reported signs and symptoms of influenza were tested using nasal pharyngeal swabs, with secretions cultured using susceptible tissue culture cell lines. Positive cultures were confirmed as influenza using immunofluorescence techniques with influenza strain specific antibodies.
Time Frame: Month 4 through Month 10 post-vaccination 1
Population: Influenza signs and symptoms were assessed in participants who had no detectable anti-M2e antibodies on Day 0, received injections on Days 0 and 30, completed the Day 60 visit, and had antibody assessments on Day 60, Per-Protocol Population.
Measure: Number; unit: Participants
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
Participants
  Signs and Symptoms of Influenza | 3 | 2 | 1 | 0
  Culture Confirmed Influenza | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Seroconversion to M2e Antigen During Initial Treatment and Follow Up Period After Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine
Description: Seroconversion was defined as an end point anti M2e antibody titer ≥ 100. Antibody responses were assessed by means of enzyme linked immunosorbent assay (ELISA)
Time Frame: Day 15 through Month 10 Post-vaccination 1
Population: Seroconversion to M2e antigen was assessed participants who had no detectable anti-M2e antibodies on Day 0, received injections on Days 0 and 30, completed the Day 60 visit, and had antibody assessments on Day 60, Per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
Participants
  Day 15 (N = 19, 20, 14, 18) | 0 | 12 | 2 | 0
  Day 30 (N = 19, 20, 14, 18) | 0 | 9 | 2 | 0
  Day 45 (N = 19, 20, 14, 18) | 6 | 19 | 9 | 1
  Day 60 (N = 19, 20, 14, 18) | 7 | 18 | 6 | 0
  Month 4 (N = 19, 20, 13, 18) | 4 | 16 | 5 | 1
  Month 10 (N = 19, 19, 12, 15) | 0 | 8 | 2 | 0

6. Primary Outcome: Geometric Mean Titers (GMTs) of Vaccine Antibodies After Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or a Placebo Vaccine.
Description: Antibody responses to the respective vaccines were assessed by means of enzyme linked immunosorbent assay (ELISA).
  A GMT value of 50.0 indicates a titer at or below the lowest limit of quantitation (LLOQ)
Time Frame: Day 15 through Month 10 Post-vaccination 1
Population: Geometric mean titers of the respective vaccine antibodies were assessed in participants who had no detectable anti-M2e antibodies on Day 0, received injections on Days 0 and 30, completed the Day 60 visit, and had antibody assessments on Day 60, Per-protocol population; per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution (1/dil)
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
1/dilution (1/dil)
  Day 15 (N = 19, 21, 14, 18) | 50.0 [50.0 to 50.0] | 200.0 [89.1 to 448.9] | 67.3 [39.3 to 115.2] | 50.0 [50.0 to 50.0]
  Day 30 (N = 19, 21, 14, 18) | 50.0 [50.0 to 50.0] | 146.4 [72.0 to 297.7] | 67.3 [39.3 to 115.2] | 50.0 [50.0 to 50.0]
  Day 45 (N = 19, 21, 14, 18) | 124.5 [57.5 to 269.4] | 887.7 [440.7 to 1788.1] | 148.6 [71.5 to 308.8] | 54.0 [45.9 to 63.5]
  Day 60 (N = 19, 21, 14, 18) | 103.7 [57.2 to 187.9] | 492.5 [241.0 to 1006.3] | 110.4 [53.0 to 230.0] | 50.0 [50.0 to 50.0]
  Month 4 (N = 19, 20, 13, 18) | 77.5 [48.8 to 123.0] | 273.2 [148.6 to 502.3] | 89.9 [48.7 to 165.9] | 52.0 [47.9 to 56.4]
  Month 10 (N = 19, 19, 12, 15) | 50.0 [50.0 to 50.0] | 100.0 [64.1 to 156.1] | 70.7 [42.3 to 118.3] | 50.0 [50.0 to 50.0]

7. Secondary Outcome: Number of Participants With Seroconversion to M2e Antigen by Immunoglobulin G (IgG) Subclasses Before and Post-Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Description: Seroconversion was defined as an antibody Titer ≥ 100. Antibody responses were assessed by means of enzyme linked immunosorbent assay (ELISA)
Time Frame: Day 0 and Day 60 Post-vaccination 1
Population: Seroconversion to M2e antigens were assessed in participants who had no detectable anti-M2e antibodies on Day 0, received injections on Days 0 and 30, completed the Day 60 visit, and had antibody assessments on Day 60, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
Participants
  IgG1 (Day 0) | 0 | 0 | 0 | 0
  IgG1 (Day 60) | 4 | 9 | 2 | 0
  IgG2 (Day 0) | 1 | 0 | 0 | 0
  IgG2 (Day 60) | 2 | 1 | 1 | 0
  IgG3 (Day 0) | 1 | 1 | 1 | 1
  IgG3 (Day 60) | 5 | 12 | 4 | 0
  IgG4 (Day 0) | 0 | 1 | 1 | 1
  IgG4 (Day 60) | 1 | 2 | 3 | 3

8. Secondary Outcome: Geometric Mean Titers of Anti-M2e Antigen by Immunoglobulin G (IgG) Subclasses Before and Post-Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Description: Antibody responses were assessed by means of enzyme linked immunosorbent assay (ELISA).
  A GMT value of 50.0 indicates a titer at or below the lowest limit of quantitation (LLOQ).
Time Frame: Day 0 and Day 60 Post-vaccination 1
Population: Geometric mean titers (GMTs) and GMT ratios of Anti-M2e antigen were assessed in participants who had no detectable anti-M2e antibodies on Day 0, received injections on Days 0 and 30, completed the Day 60 visit, and had antibody assessments on Day 60, per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution (1/dil)
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
1/dilution (1/dil)
  IgG1 (Day 0) | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  IgG1 (Day 60) | 73.5 [44.8 to 121] | 135 [74.8 to 242] | 65.8 [40.4 to 107] | 50.0 [50.0 to 50.0]
  IgG2 (Day 0) | 53.2 [46.7 to 60.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  IgG2 (Day 60) | 56.2 [47.1 to 67.0] | 57.0 [43.4 to 74.8] | 56.2 [43.7 to 72.4] | 50.0 [50.0 to 50.0]
  IgG3 (Day 0) | 54.7 [45.2 to 66.2] | 54.4 [45.6 to 65.0] | 56.3 [43.5 to 72.9] | 52.2 [47.6 to 57.3]
  IgG3 (Day 60) | 113 [55.7 to 228] | 233 [111 to 488] | 84.3 [48.9 to 145] | 50.0 [50.0 to 50.0]
  IgG4 (Day 0) | 50.0 [50.0 to 50.0] | 51.8 [48.1 to 55.8] | 52.6 [47.2 to 58.6] | 52.0 [47.9 to 56.5]
  IgG4 (Day 60) | 52.3 [47.6 to 57.4] | 55.5 [47.4 to 65.1] | 68.8 [46.5 to 102] | 63.5 [47.1 to 85.5]

9. Secondary Outcome: Geometric Mean Titer Ratios of Anti-M2e Antigen by Immunoglobulin G (IgG) Subclasses Before and Post-Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Description: Antibody responses were assessed by means of enzyme linked immunosorbent assay (ELISA).
Time Frame: Day 0 and Day 60 Post-vaccination 1
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
Ratio
  GMT Ratio (Day 60/Day 0) | 1.47 [0.896 to 2.41] | 2.69 [1.50 to 4.84] | 1.32 [0.809 to 2.14] | 1 [1.0 to 1.0]
  GMT Ratio (Day 60/Day 0) | 1.06 [0.964 to 1.16] | 1.14 [0.867 to 1.50] | 1.12 [0.873 to 1.45] | 1.0 [1.0 to 1.0]
  GMT Ratio (Day 60/Day 0) | 2.06 [0.969 to 4.34] | 4.28 [2.03 to 9.02] | 1.50 [1.00 to 2.23] | 0.957 [0.873 to 1.05]
  GMT Ratio (Day 60/Day 0) | 1.05 [0.952 to 1.15] | 1.07 [0.895 to 1.28] | 1.31 [0.948 to 1.80] | 1.22 [0.910 to 1.64]

10. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-Hepatitis B Core Antibodies Using Immunoglobulin G (IgG) ELISA Before and Post-Vaccination With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Description: Antibody responses were assessed by means of enzyme linked immunosorbent assay (ELISA)
Time Frame: Day 0 and Day 15 through Month 10 post-vaccination 1
Population: Antibody responses were assessed in participants who had no detectable anti-M2e antibodies on Day 0, received injections on Days 0 and 30, completed the Day 60 visit, and had antibody assessments on Day 60, Per-Protocol Population.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/diultion (1/dil)
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
1/diultion (1/dil)
  Day 0 (N = 19, 20, 14, 18) | 63.9 [50.0 to 81.6] | 53.0 [46.9 to 60.0] | 58.2 [46.5 to 72.7] | 66.9 [45.2 to 98.9]
  Day 15 (N = 19, 20, 14, 18) | 367 [214 to 630] | 1779 [1216 to 2601] | 232 [124 to 435] | 65.8 [45.3 to 95.6]
  Day 30 (N = 19, 20, 14, 18) | 312 [179 to 542] | 1239 [831 to 1847] | 161 [87.5 to 298] | 66.0 [44.9 to 97.0]
  Day 45 (N = 19, 20, 14, 18) | 2353 [1328 to 4168] | 13402 [9434 to 19040] | 794 [405 to 1555] | 68.0 [45.1 to 102]
  Day 60 (N = 19, 20, 14, 18) | 2028 [1191 to 3453] | 10359 [6778 to 15833] | 637 [312 to 1301] | 64.2 [42.3 to 97.3]
  Month 4 (N = 19, 20, 13, 18) | 1387 [834 to 2307] | 7936 [5294 to 11896] | 517 [219 to 1218] | 59.6 [41.1 to 86.5]
  Month 10 (N = 19, 19, 12, 15) | 311 [197 to 489] | 2110 [1235 to 3607] | 244 [95.4 to 623] | 65.6 [41.7 to 103]

11. Secondary Outcome: Number of Participants With Seropositivity to Hepatitis B Core Antigen Pre- and Post-Vaccination 1 With ACAM FLU A, or ACAM FLU A With Adjuvant, or Placebo Vaccine.
Description: Seropositivity with ELISA was defined as a Pre- or post-vaccination antibody titer ≥ 100. Seropositivity with the Commercial Kit method was defined as a positive pre- or post-vaccination response.
  Seropositivity were assessed by means of enzyme linked immunosorbent assay (ELISA) and the Commercial Kit methods
Time Frame: Day 0 and Day 15 through Month 10 Post-vaccination 1
Population: Seropositivity to Hepatitis B core antigen was assessed in participants who had no detectable anti-M2e antibodies on Day 0, received injections on Days 0 and 30, completed the Day 60 visit, and had antibody assessments on Day 60, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Number analyzed (Participants) | 19 | 20 | 14 | 18
Participants
  ELISA Day 0 (N = 19, 20, 14, 18) | 4 | 1 | 2 | 3
  ELISA Day 15 (N = 19, 20, 14, 18) | 17 | 20 | 11 | 3
  ELISA Day 30 (N = 19, 20, 14, 18) | 17 | 20 | 9 | 3
  ELISA Day 45 (N = 19, 20, 14, 18) | 19 | 20 | 14 | 3
  ELISA Day 60 (N = 19, 20, 14, 18) | 19 | 20 | 14 | 2
  ELISA Month 4 (N = 19, 20, 13, 18) | 19 | 20 | 12 | 1
  ELISA Month 10 (N = 19, 19, 12, 15) | 17 | 19 | 8 | 2
  Commercial Kit Day 0 (N = 19, 20, 14, 18) | 0 | 0 | 0 | 0
  Commercial Kit Day 60 (N = 19, 19, 13, 18) | 19 | 19 | 12 | 0
  Commercial Kit Month 10 (N = 19, 19, 12, 15) | 15 | 19 | 9 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) up to 9 months post-vaccination 1
Arm/Group | ACAM-FLU-A Adjuvanted With Alhydrogel | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 | ACAM FLU A Without Adjuvant | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/23 | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 22/22 | 23/23 | 20/21 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACAM-FLU-A Adjuvanted With Alhydrogel (N=22) | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 (N=23) | ACAM FLU A Without Adjuvant (N=21) | Saline Placebo (N=21)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACAM-FLU-A Adjuvanted With Alhydrogel (N=22) | ACAM-FLU-A Adjuvanted With Stimulon® QS-21 (N=23) | ACAM FLU A Without Adjuvant (N=21) | Saline Placebo (N=21)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Chills (General disorders) | 0 | 9 | 0 | 2
Fatigue (General disorders) | 5 | 12 | 3 | 5
Injection site erythema (General disorders) | 3 | 7 | 4 | 2
Injection site induration (General disorders) | 2 | 0 | 3 | 0
Injection site pain (General disorders) | 20 | 20 | 16 | 4
Injection site pruritus (General disorders) | 0 | 3 | 0 | 2
Injection site swelling (General disorders) | 3 | 8 | 0 | 0
Malaise (General disorders) | 2 | 9 | 2 | 2
Pyrexia (General disorders) | 4 | 10 | 4 | 2
Alanine aminotransferase increase (Investigations) | 0 | 2 | 2 | 0
Aspartate aminotransferase increase (Investigations) | 0 | 3 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 0 | 2
Blood creatinine increased (Investigations) | 2 | 0 | 3 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 2
Blood potassium increased (Investigations) | 2 | 0 | 3 | 0
Haemoglobin decreased (Investigations) | 4 | 6 | 5 | 5
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 0
White blood cell count increased (Investigations) | 0 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 12 | 6 | 3
Headache (Nervous system disorders) | 6 | 9 | 5 | 2
Syncope vasovagal (Nervous system disorders) | 0 | 2 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.